CLINICAL TRIAL: NCT02353221
Title: California Pacific Medical Center Early Undifferentiated Arthritis Registry
Brief Title: CPMC Early Undifferentiated Arthritis Registry
Acronym: CEUAR
Status: Completed | Type: Observational
Sponsor: California Pacific Medical Center Research Institute (Other)
Responsible Party: Principal Investigator, Pedro Ruiz, Rheumatologist, California Pacific Medical Center Research Institute
Other Study IDs: GRO
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Early Undifferentiated Arthritis
Keywords: Early arthritis; undiferentiated arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Blood samples: Our objective is to create a repository that includes PBMCs and serum samples suitable for functional assays as well as nucleic acid analysis. These efforts will make our cohort a unique source to measure PBMC antigen-specific proliferation, cytokine and chemokine secretion, and activation markers expression among others. Blood will be fractionated for serum analysis and cell analysis. PBMCs will be sorted into neutrophils, B cells, T cells, and monocytes. Cells will be used for RNA and DNA extraction and analysis, for functional assays involving cytokine and chemokine production, cell proliferation, and expression of surface markers of activation.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects: Entry criteria include being at least 18 years old at screening visit, being able to understand the information given to them and to give written informed consent, willingness to comply with the requirements of the data collection, absence of a diagnose of autoimmune disease or inflammatory arthritis, and absence of a previous treatment with any disease modifying anti-rheumatic drug (DMARD). We will exclude patients that are pregnant or intend to become pregnant during the time of follow up.
- Controls: Healthy control subjects will be recruited based on similar criteria as study subjects. Our effort will be to include age and gender matched control subjects in the registry. We will be also aiming to match environmental characteristics (i.e. partners living in same location as registry subject or in a radius of 10 miles for at least one year previous to the date of evaluation) or genetic background (i.e. by asking the participation of first-degree relatives)

SUMMARY:
The CPMC early arthritis registry will recruit participants from a population of new patients undergoing evaluation at the office of participating physicians. Patients enrolled in the registry will undergo longitudinal observation and sampling. The investigators will collect questionnaire data and create a biological sample repository. The information obtained will be use to generate hypotheses aimed at explaining how environmental and genetic factors are interrelated to influence UA disease outcomes. Analysis will be performed on the patient's data and biological samples in order to; A. Assess the epidemiological and clinical characteristics of patients with early arthritis in the referral pool at CPMC.

B. Analyze the phenotype and genotype of peripheral blood mononuclear cells (PBMC) from individual patients based on their chemokine/cytokine secretion, cell adhesion molecule expression, gene expression, DNA methylation and non coding RNA profiles.

C. Generate hypothesis aimed to identify clinical criteria and novel biomarkers to be used in the diagnosis, prognosis, and therapeutic decisions for patients with early UA

DETAILED DESCRIPTION:
Experimental Design/Procedural Methods:

Study Objectives:

The CPMC early arthritis registry will recruit participants from a population of new patients undergoing evaluation at the office of participating physicians. Patients enrolled in the registry will undergo longitudinal observation and sampling. The investigators will collect questionnaire data and create a biological sample repository. The information obtained will be use to generate hypotheses aimed at explaining how environmental and genetic factors are interrelated to influence UA disease outcomes. Analysis will be performed on the patient's data and biological samples in order to; A. Assess the epidemiological and clinical characteristics of patients with early arthritis in the referral pool at CPMC.

B. Analyze the phenotype and genotype of peripheral blood mononuclear cells (PBMC) from individual patients based on their chemokine/cytokine secretion, cell adhesion molecule expression, gene expression, DNA methylation and non coding RNA profiles.

C. Generate hypothesis aimed to identify clinical criteria and novel biomarkers to be used in the diagnosis, prognosis, and therapeutic decisions for patients with early UA.

Design:

A. Prospective longitudinal registry. B. Participants: Any patient undergoing evaluation for arthritis will be considered eligible. The pool of potential subjects will include any patient presenting to the office of participating physicians for evaluation of arthritis. As an estimate, Pacific Rheumatology Associates, our private practice office in San Francisco, performed approximately 1000 consultations in 2013 on undiagnosed arthritis.

C. Entry criteria include being at least 18 years old at screening visit, being able to understand the information given to them and to give written informed consent, willingness to comply with the requirements of the data collection, absence of a diagnose of autoimmune disease or inflammatory arthritis, and absence of a previous treatment with any disease modifying anti-rheumatic drug (DMARD). We will exclude patients that are pregnant or intend to become pregnant during the time of follow up.

Healthy control subjects will be recruited based on similar criteria as study subjects. Our effort will be to include age and gender matched control subjects in the registry. We will be also aiming to match environmental characteristics (i.e. partners living in same location as registry subject or in a radius of 10 miles for at least one year previous to the date of evaluation) or genetic background (i.e. by asking the participation of first-degree relatives).

D. Measurements:

i. Demographics, clinical, and environmental characteristics: Patients and controls will fill out an epidemiological survey of the main demographic characteristics (i.e. age, gender, ethnicity, etc), clinical characteristics (i.e. past medical history, family history, medication allergies, and medications) and environmental characteristics (socio-economic status, sleep habits, tobacco exposure, diet, etc.) ii. Outcomes: 1. A Health Assessment Questionnaire (HAQ) 6, a Sleep Questionnaire 7, and a semi quantitative food frequency questionnaire 8 will be applied at the date of initial evaluation to patients and controls. These questionnaires will be administered again once a participant considers her/his symptoms had improved or she/he had failed the initial therapeutic intervention. At this point we will also be including the appropriate control subject in the sampling. Patients will have a DAS28 score calculated by a physician during each medical evaluation.

2. Patient's follow up either by personal or phone interview after initial visit will be at six, 12, and 24 months in order to record any definitive diagnosis of inflammatory arthritis.

3. A participant will be requested to provide a blood sample at the initial evaluation visit and/or during an active disease phase if there is no disease activity on the first office visit. Another blood sample will be collected after the initial therapeutic intervention regardless of whether there is inactive or low activity disease phase as per patient's subjective assessment.

Follow up interviews whenever requiring a personal visit will be conducted at the office of participating physicians.

iii. Blood samples: Our objective is to create a repository that includes PBMCs and serum samples suitable for functional assays as well as nucleic acid analysis. These efforts will make our cohort a unique source to measure PBMC antigen-specific proliferation, cytokine and chemokine secretion, and activation markers expression among others. As described above, participants will be ask to donate a blood sample on a period of disease activity and a period of disease inactivity or low activity as calculated by their DAS28 scores. Blood will be fractionated for serum analysis and cell analysis. PBMCs will be sorted into neutrophils, B cells, T cells, and monocytes. Cells will be used for RNA and DNA extraction and analysis, for functional assays involving cytokine and chemokine production, cell proliferation, and expression of surface markers of activation. Serum and cells will be stored at the CPMC Research Institute. Serum samples stored at -70° C will be used for soluble cytokine and chemokine analysis. Sorted cells will be collected in RNA-preserving media and stored in liquid nitrogen and used for nucleic acid analysis (mRNA, small RNA, cDNA, genomic DNA). An additional sample of PBMCs will be collected in dimethyl sulfoxide (DMSO) and stored in liquid nitrogen to be used for functional assays including cell proliferation and activation markers expression.

iv. Imaging: We will request a copy of any radiological assessment related with the patient work up for diagnosis and evaluation of the arthritis. We will be also registering any imaging studies related to follow up visits.

E. HIPAA and Informed Consent:

Patients eligible will be invited to enroll in the registry and informed consent will be obtained. Patients will be provided with a detailed description of the aims, expectations, and possible complications related to the participation in the study. Participation will be completely voluntary. The project will strictly abide by the Health Insurance and Accountability Act (HIPAA) and the California Confidentiality of Medical Information Act and will be subjected to the approval by the California Pacific Medical Center Institutional Review Board.

ELIGIBILITY:
Inclusion Criteria:

* Entry criteria include being at least 18 years old at screening visit
* Being able to understand the information given to them and to give written informed consent
* Willingness to comply with the requirements of the data collection
* Absence of a diagnose of autoimmune disease or inflammatory arthritis
* Absence of a previous treatment with any disease modifying anti-rheumatic drug (DMARD)

Exclusion Criteria:

* We will exclude patients that are pregnant or intend to become pregnant during the time of follow up.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants: Any patient undergoing evaluation for arthritis will be considered eligible. The pool of potential subjects will include any patient presenting to the office of participating physicians for evaluation of arthritis.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2015-01; Primary Completion 2022-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Diagnosis of inflammatory arthritis | one year

CONTACTS AND LOCATIONS:
Overall Officials: Pedro J. Ruiz, MD PhD, Principal Investigator — CPMCRI
Locations (1):
- California Pacific Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Hitchon CA, Peschken CA, Shaikh S, El-Gabalawy HS. Early undifferentiated arthritis. Rheum Dis Clin North Am 2005;31:605-26. 2. Kremer JM, Gibofsky A, Greenberg JD. The role of drug and disease registries in rheumatic disease epidemiology. Curr Opin Rheumatol 2008;20:123-30. 3. Pincus T. Limitations of randomized clinical trials in chronic diseases: explanations and recommendations. Adv Mind Body Med 2002;18:14-21. 4. Goekoop-Ruiterman YP, de Vries-Bouwstra JK, Allaart CF, et al. Clinical and radiographic outcomes of four different treatment strategies in patients with early rheumatoid arthritis (the BeSt study): a randomized, controlled trial. Arthritis Rheum 2005;52:3381-90. 5. Lard LR, Visser H, Speyer I, et al. Early versus delayed treatment in patients with recent-onset rheumatoid arthritis: comparison of two cohorts who received different treatment strategies. Am J Med 2001;111:446-51. 6. Lillegraven S, Kvien TK. Measuring disability and quality of life in established rheumatoid arthritis. Best Pract Res Clin Rheumatol 2007;21:827-40. 7. Yeboah J, Redline S, Johnson C, et al. Association between sleep apnea, snoring, incident cardiovascular events and all-cause mortality in an adult population: MESA. Atherosclerosis 2011;219:963-8. 8. Willett WC, Sampson L, Stampfer MJ, et al. Reproducibility and validity of a semiquantitative food frequency questionnaire. American journal of epidemiology 1985;122:51-65.